CLINICAL TRIAL: NCT02701803
Title: Ambulatory Movement Registration in Patients With Deep Brain Stimulation and Continuous Intraduodenal Levodopa Therapy
Brief Title: Parkinson's KinetiGraph, PKG in Patients With Deep Brain Stimulation and Continuous Levodopa Infusion Therapy
Status: Completed | Type: Observational
Sponsor: Hospital District of Helsinki and Uusimaa (Other)
Responsible Party: Principal Investigator, Maija Koivu, Specialising physician, Hospital District of Helsinki and Uusimaa
Other Study IDs: HospitalDHU
Record Dates: First submitted 2016-02-12; First posted 2016-03-08 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Parkinson's KinetiGraph™ logger — Logger is recording device which records the movement and acceleration of upper extremity

SUMMARY:
In this study the aim is to evaluate the outcome of deep brain stimulation (DBS) and continuous intraduodenal levodopa therapy in patients with advanced Parkinson' disease by using Parkinson's KinetiGraph™ device which is a movement and acceleration measuring device. In this study we also evaluate the usability of Parkinson's KinetiGraph™ device by comparing it with written patient diaries.

DETAILED DESCRIPTION:
In this study the aim is to evaluate the outcome of deep brain stimulation (DBS) and continuous intraduodenal levodopa therapy in patients with advanced Parkinson' disease by using Parkinson's KinetiGraph™ logger (PKG) device which is a movement and acceleration measuring device.

A measurement is done before and after the implantation of selected therapy. PKG will measure automatically in every two minutes the movement of selected limb (usually the more affected upper extremity) for six days. At the same time a patient will keep a written diary of his/her Parkinsonian symptoms. Diary and collected PKG data will be compared. PKG will also remind with vibration the patient of the time drug administration and the patient can confirm this with pressing a button on PKG. The collected data will be transmitted to a computer and analyzed mathematically to produce a visual graph of daily movements. The aim is to evaluate PKG's usability in measuring Parkinsonian symptoms and in evaluation the outcome of DBS and levodopa therapy. Main parameters in evaluation are bradykinesia score and dyskinesia score.

ELIGIBILITY:
Inclusion Criteria:

* Patient with diagnosed Parkinson's disease
* Parkinson's disease is in advanced state (defined by the treating physician)
* A good response with over 30 % improvement of scores in Unified Parkinson's disease rating scale part III in pre-DBS evaluation

Exclusion Criteria:

* Age older than 70 years (this is a clinical exclusion criteria for DBS treatment)
* No history of psychosis or depression (this is a clinical exclusion criteria for DBS and intraduodenal levodopa therapy)
* No diagnosed dementia (this is a clinical exclusion criteria for DBS and intraduodenal levodopa therapy)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population is consisted of patients with advanced Parkinson's disease in HUH neurological clinic. The treatment decision of deep brain stimulation and/or continuous intraduodenal levodopa therapy is done clinically by the treating physician. The patients are enrolled in the study after the clinical decision is made.
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2015-10; Primary Completion 2017-12 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Bradykinesia score | 6 months
  BKS is summary of bradykinesia presented in PKG recordings, BKS, 0 - 50

SECONDARY OUTCOMES:
Dyskinesia score | 6 months
  DKS summary of dyskinesia presented in PKG recordings, DKS, 0 - 50

CONTACTS AND LOCATIONS:
Overall Officials: Eero Pekkonen, M.D., Ph.D., Study Director — HUH, Meilahti Hospital, department of neurology
Locations (1):
- HUH Meilahti Hospital, department of neurology, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No